CLINICAL TRIAL: NCT00158171
Title: Interventions for Tobacco Dependent Adolescents
Brief Title: Effectiveness of Various Smoking Cessation Therapies in Reducing Smoking in Adolescents - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Dorothy Hatsukami, UMN
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-14538-1; R01-14538-1; DPMC
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-10

CONDITIONS: Smoking Cessation; Tobacco Use Disorder
Keywords: smoking addiction
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — Nicotine Replacement Therapy; Nicotine Chewing Gum; Tobacco Use Cessation Devices; Nicotine; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Nicotine patch
  Interventions: Drug: Nicotine Replacement Therapies
- 2 (Experimental): Nicotine gum
  Interventions: Drug: Nicotine patch
- 3 (Placebo Comparator): Folic acid
  Interventions: Dietary Supplement: Folic Acid

INTERVENTIONS:
Drug: Nicotine Replacement Therapies — Nicotine gum 2 & 4 mg dependent on baseline smoking rate
  Other Names: Nicorette
  Arms: 1
Drug: Nicotine patch — 21, 14 or 7 mg patch dependent on baseline smoking rate
  Other Names: Nicoderm
  Arms: 2
Dietary Supplement: Folic Acid — 400 mg
  Arms: 3

SUMMARY:
Currently one in five high school students smokes. Smoking can harm adolescents well before they reach adulthood by causing a number of immediate, sometimes irreversible, health risks and problems. This study will compare the effectiveness of treatment with bupropion, a nicotine patch, or nicotine gum in supporting the reduction of smoking in adolescent smokers.

DETAILED DESCRIPTION:
Among adolescents, the short-term health effects of smoking include damage to the respiratory system, addiction to nicotine, and the associated risk of other drug use. Adolescents are at greater risk for long-term health problems because most young people who smoke regularly continue to smoke throughout adulthood. This study will compare the effectiveness of treatment with bupropion, a nicotine patch, or nicotine gum in supporting the reduction of smoking in adolescent smokers. The study will also assess whether reduction of smoking leads to continued involvement in treatment, less toxic cigarette exposure, and improved motivation to quit.

This open-label study will last a total of 6 weeks. Baseline measurements will be taken twice a week at study visits for the first two weeks to assess vital signs and smoking behavior. Participants will aslo use a computerized device outside of study visits to monitor their own smoking habits. At Week 3, participants will be randomly assigned to receive bupropion, a nicotine patch, nicotine gum, or placebo. Participants will be asked to limit the frequency of their smoking to 75% of what it was during baseline. During Weeks 4, 5, and 6, participants will be expected to reduce smoking behavior to 50% of what it was at baseline. Customized doses of nicotine patches and nicotine gum, relative to the amount of cigarettes a participant smoked during baseline, will be dispensed weekly. Participants receiving bupropion or placebo will receive medication at each study visit and will take one pill daily. During treatment, study visits will occur once weekly. At each study visit, all participants will receive a 10- to 15-minute standardized behavioral therapy session aimed at supporting smoking reduction. Smoking habits and vital signs will be assessed and the effects of the treatments will be determined. There will be one follow-up visit 3 months post-intervention, at which time smoking status will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months of daily cigarette smoking
* No use of other tobacco products
* Motivated to reduce or quit smoking
* Not currently using medications to quit smoking
* Agree to use an effective form of contraception throughout the study

Exclusion Criteria:

* People for whom use of nicotine replacement therapy or bupropion is medically inadvisable
* History of alcohol or drug abuse within 6 months of enrollment
* History of emotional problems (as assessed by the Adolescent Symptoms Inventory) within 6 months prior to enrollment
* Currently on an unstable dose of psychoactive medications
* Currently taking medications that may react with one of the treatment medications
* Pregnant

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 128 (Actual)
Dates: Start 2002-04; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Reduction in tobacco toxicant exposure | Weeks 2, 5 and 17

SECONDARY OUTCOMES:
Motivation and self-efficacy to quit; measured at Weeks 5 and 17 | Weeks 5 and 17
Reduction in cigarettes per day | Weeks 5 and 17
Smoking cessation | Weeks 5 and 17

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States